CLINICAL TRIAL: NCT00654160
Title: A Pharmacogenetic-Based Phase I Trial of Irinotecan, 5-Fluorouracil, and Leucovorin (FOLFIRI) in Patients With Advanced Gastrointestinal Cancer
Brief Title: Irinotecan, Fluorouracil, and Leucovorin in Treating Patients With Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000592931; P30CA015083 (NIH); MC064G (Other: Mayo Clinic Cancer Center); NCI-2009-01216 (Registry Identifier: CTRP)
Record Dates: First submitted 2008-04-04; First posted 2008-04-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2016-09

CONDITIONS: Anal Cancer; Carcinoma of the Appendix; Colorectal Cancer; Esophageal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Gastrointestinal Carcinoid Tumor; Gastrointestinal Stromal Tumor; Liver Cancer; Pancreatic Cancer; Small Intestine Cancer
Keywords: stage IIIB anal cancer; stage IV anal cancer; recurrent anal cancer; carcinoma of the appendix; stage III colon cancer; stage IV colon cancer; recurrent colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrointestinal stromal tumor; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; recurrent small intestine cancer; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma
MeSH Terms: conditions — Anus Neoplasms; Appendiceal Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Liver Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular | interventions — Fluorouracil; Irinotecan; Leucovorin; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Other: pharmacogenomic studies
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan when given together with fluorouracil and leucovorin in treating patients with advanced gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of irinotecan hydrochloride in FOLFIRI for each respective UGT1A1 TA indel genotype grouping (group 1 [7/7, 7/8, 8/8], group 2 [6/7, 5/7, 5/8 ,6/8], and group 3 [6/6, 5/6, 5/5]).

Secondary

* Determine the molecular basis of toxicity, other than UGT1A1 variants, in FOLFIRI-treated cancer patients.
* Determine the pharmacodynamic molecular profiles of cell signaling pathways associated with the development and severity of early and late specific toxicities in cancer patients treated with FOLFIRI.

OUTLINE: This is a dose-escalation study of irinotecan hydrochloride. Patients are stratified according to genotype of UGT1A1 TA indel.

* Group 1 ( TA genotype 7/7, 7/8, 8/8): Patients receive irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV bolus over 5 minutes followed by IV continuously over 46 hours on days 1-3.
* Group 2 (TA genotype 6/7, 6/7, 5/8, 6/8): Patients receive treatment as in group 1 with a higher initial dose of irinotecan hydrochloride.
* Group 3 (TA genotype 5/5, 5/6, 6/6): Patients receive treatment as in group 2. In all groups, treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and periodically during study for pharmacokinetics, dihydropyridine deaminase enzyme assay, and pathway expression analysis.

After completion of study treatment, patients are followed every 6 weeks for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed diagnosis of gastrointestinal cancer

  * Advanced, unresectable disease
* Confirmation of UGT1A1 TA indel genotype
* Measurable or evaluable (non-measurable) disease

  * Measurable disease is defined as ≥ 1 lesion that can be accurately measured (longest diameter to be recorded) as ≥ 2.0 cm with conventional techniques or as ≥ 1.0 cm with spiral CT scan

    * Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules, palpable lymph nodes)
    * Lesions on chest x-ray are acceptable as measurable lesions when they are clearly defined and surrounded by aerated lung
  * The following are considered non-measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusions
    * Lymphangitis cutis/ pulmonis
    * Inflammatory breast disease
    * Abdominal masses (not followed by CR scan or MRI)
    * Cystic lesions
    * All other lesions (or sites of disease), including small lesions (longest diameter < 2.0 cm with conventional techniques or as < 1.0 cm with spiral CT)
* No known central nervous system metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Inclusion criteria

* Life expectancy ≥ 12 weeks.
* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* SGOT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN if liver metastases)
* Total Bilirubin ≤ ULN for patients in group 3 and ≤ 2.0 times ULN for patients in groups 1 and 2
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for the duration of study treatment
* Willing to provide blood samples for mandatory translational studies

Exclusion criteria

* Known allergy to irinotecan hydrochloride-related agents (e.g., topotecan), 5-fluorouracil, and/or leucovorin calcium
* Active or uncontrolled infection
* Evidence of serious intercurrent illness (e.g., unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia)

PRIOR CONCURRENT THERAPY:

* Recovered from all toxicities
* More than 4 weeks since prior major surgery
* More than 2 weeks since completion of prior radiotherapy

  * No prior radiotherapy to > 25% of bone marrow
* More than 2 week since prior cytotoxic chemotherapy, biologic therapy, or immunotherapy
* No concurrent sargramostim (GM-CSF)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2012-12-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of genotype-based dosing of FOLFIRI with or without monoclonal antibody therapy

SECONDARY OUTCOMES:
Response rate of genotype-based dosing in the subset of patients that has colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Robert McWilliams, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States